CLINICAL TRIAL: NCT06570304
Title: Prevention of Retained Items iN Childbirth Environment and Surgical Sites- Clinical Usability Study
Brief Title: Prevention of Retained Items iN Childbirth Environment and Surgical Sites
Acronym: PRINCESS
Status: Not yet recruiting | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Collaborators: Innovate UK (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024SUR130
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Retained Surgical Items
MeSH Terms: conditions — Foreign Bodies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- iCount Device: A novel external device which can count the swabs and surgical tampons used during childbirth in an objective and validated manner.
  Interventions: Procedure: iCount Device
- User Feedback Survey: Anonymised feedback data will be collected from 20 staff users about the user experience and usability of the device. This will be conducted with an online survey questionnaire designed with advice from ergonomics experts after an extensive literature review of human factors-ergonomics principles and MHRA guidance about conducting medical device usability
  5 staff users will be randomly selected from the consent forms to have semi-structured interviews developed in accordance with qualitative research methodology for medical device usability testing and user experience.

INTERVENTIONS:
Procedure: iCount Device — Designed as single use. Intended purpose - To be used to count swabs and tampons after surgery in an objective manner. This is intended to be used in patients during and just after surgery.
  This is a device accessory.
  Groups: iCount Device

SUMMARY:
To evaluate the user confidence in the confirmation of correct counts using a novel device and to assess clinical usability of the device during surgery.

DETAILED DESCRIPTION:
Accidentally retained surgical items or swabs are well-recognised errors that result in adverse consequences for patients. This error is one of the commonest "Never Events" - patient safety incidents that are considered preventable. Although uncommon, these incidents can have devastating consequences. Retained surgical items have 70% re-interventions, reaching 80% morbidity and 35% mortality. (Birolini et al, 2016) 1

Swabs or sponges are like small towels that soak up blood and body fluids so that the surgeon can visualise the operating area effectively. Swabs are used in all areas of surgery which include operations on the tummy, chest, limbs. They are also used in the vagina during childbirth, to assess for tears and to minimise blood oozing from the vagina.

The common risk factors for this error are out of hours surgical or childbirth procedures, multiple handovers in the care of the patient, raised BMI (Body Mass Index) and unplanned change to the operative intervention. (Gawande et al, 2003)2 As the name suggests, a 'never event' should never happen. Unfortunately, incidents involving surgical swabs being left behind, particularly during a caesarean section or a perineal repair following a vaginal birth, are still happening despite over 100 years of institutional awareness of the problem and tentative solutions being implemented in clinical practice.

Never-events involving retained surgical swabs are a widespread problem affecting healthcare systems worldwide. It is therefore reasonable to ask the question: why are surgical swabs being left behind and what can be done to prevent this from happening?

Patient safety is a well-known priority for the European commission, WHO and the NHS. Some of the National/International reports highlighting this problem:

* CQC-Opening the door to change (2018)
* US Joint Commission report: Preventing unintended retained foreign objects (2019)
* The Australian Commission on Safety and Quality in Health Care and The New Zealand Health Quality and Safety Commission (2015)
* Healthcare Safety Investigation Branch (HSIB,UK) investigation I2018/025 (2019)

ELIGIBILITY:
Inclusion Criteria:

1. Patients due to undergo surgery at the chosen NHS Trust.
2. Patients 18 years or older and consented to participation after an informed choice.

Exclusion Criteria:

1. Under 18 years of age
2. Emergency surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be pregnant women during labour.
  Staff who work in the operating theatres and are involved in performing swab and instrument counts. Consented to participation after an informed choice.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Understanding user experience/usability factors | 12 months
  User responses on Likert scale for the various usability factors such as user confidence in the accuracy of counts, functional aspects and ease of use collected with an online software-assisted survey.
How the device sits within the current system | 12 months
  The purpose is to obtain user centred narratives and a rich qualitative data. Semi-structured interviews of staff will be conducted via a virtual platform or in a safe face-to-face manner. These will be recorded with a dictaphone recording device or Microsoft teams auto-transcription

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Desai, Principal Investigator — The Royal Wolverhampton NHS Trust